CLINICAL TRIAL: NCT02091700
Title: ObseRvation of PeripHEral rEtinal Morphology in Normal
Brief Title: ObseRvation of PeripHEral rEtinal Morphology in Normals
Acronym: ORPHEE2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Optos, PLC (Industry)
Collaborators: Medical Center Ophthalmology Associates San Antonio, Texas (Unknown)
Responsible Party: Sponsor
Other Study IDs: OPT1010
Record Dates: First submitted 2014-03-05; First posted 2014-03-19 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Healthy
Keywords: Normal; Healthy; Normal healthy patient
MeSH Terms: interventions — Indocyanine Green

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Normals: Subjects with normal visual and retinal function will be enrolled
  Interventions: Other: Indocyanine Green ICG

INTERVENTIONS:
Other: Indocyanine Green ICG

SUMMARY:
To develop a database of the peripheral choroidal circulation using ultra widefield (UWF) imaging. This database will serve as a quantitative reference tool for the comparison of subjects to a database of known normal subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects older than 20 years old with good general health.
* Subject is capable of giving consent.
* The subject is able and willing to comply with the study procedures.
* Subjects with ocular media clear enough to allow good quality ocular imaging.
* Normal subjects with no known retinal or choroidal disease.

Exclusion Criteria:

* Subjects under 20 years old.
* Subjects with contraindications to dilation.
* Subjects with a history of epilepsy.
* Subjects with a known allergy to iodine, shellfish or intra-venous x-ray contrast dyes.
* Subjects who are or who may be pregnant.
* Subjects with past history of any vitreoretinal disease or surgery such as retinal detachment, epiretinal membrane, or vitreous hemorrhage.
* Subjects with any ocular condition that interferes with good quality image acquisition, such as corneal opacities, cataract, and dense vitreous hemorrhage.
* Subjects with any evidence of any retinal or optic nerve disease including glaucoma.
* Subjects with any anterior segment disease with the exception of common ocular surface disorders (blepharitis, dry eye).
* Subjects with medical conditions that interfere with the subject's compliance to study procedures such as inability of the subject to maintain steady head or eye positioning as in patients of ataxia or nystagmus.
* Subjects with a history of Diabetes, uncontrolled blood pressure (defined as systolic >/= 160mmHg and/or diastolic >/= 90 mmHg), and Vascular Disease (cardiovascular, peripheral vascular, or cerebrovascular).
* Subjects on vasodilators.
* Subject's refusal.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal subjects with no known retinal disease or choroidal disease.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Develop a database of peripheral retinal circulation in normals using UWF-ICG imaging | 1 day

SECONDARY OUTCOMES:
Develop a database of peripheral retinal morphology on age stratified normals using color, AF and ICG imaging | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Michael Singer, MD, Principal Investigator — Medical Center Ophthalmology Associates
Locations (1):
- Medical Center Ophthalmology Associates, San Antonio, Texas, United States